CLINICAL TRIAL: NCT00496756
Title: A Phase II Study of Sorafenib in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Sorafenib in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low accrual rate
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0081-06-FB; P30CA036727 (NIH)
Record Dates: First submitted 2007-07-03; First posted 2007-07-04 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2023-10-26 (Actual); Status verified 2023-10

CONDITIONS: Kidney Cancer
Keywords: clear cell renal cell carcinoma; stage III renal cell cancer; stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sorafenib (Other): The initial dose of Sorafenib will be administered orally with a dose of 400 mg twice a day, daily. Intrapatient dose escalation will occur as defined in the table below, providing no dose limiting toxicity (Grade 3 or 4) is observed. If grade 3 or 4 toxicity is observed, delay and dose modification will occur as defined in protocol. Once dose level 3 is reached, the patient will remain at that dose as defined in following section.
  Dose Level 1 Day 1-28 400 mg b.i.d. Dose Level 2 Day 29-56 600 mg b.i.d. Dose Level 3 Day 57- 800 mg b.i.d.
  A treatment cycle will be 4 weeks.
  Two 4-week cycles will be administered. At the completion of two cycles (week 8), restaging will occur. Patients will continue on therapy per study protocol.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Sorafenib — initial dose of Sorafenib will be administered orally with a dose of 400 mg twice a day, daily.Intrapatient dose escalation will occur providing no dose limiting toxicity (Grade 3 or 4) is observed. Dose level 2 600mg. Dose level 2 800mg
  Other Names: Nexavar

SUMMARY:
RATIONALE: Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying the side effects and how well sorafenib works in treating patients with metastatic or unresectable kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the safety and toxicity of dose escalating sorafenib tosylate in patients with metastatic or unresectable renal cell carcinoma.

Secondary

* Determine tumor response in these patients.
* Determine time to progression in these patients.
* Determine overall survival of these patients.

Tertiary

* Collect data on angiogenesis inhibition induced by sorafenib tosylate.
* Collect data on immunomodulatory effects of sorafenib tosylate.

OUTLINE: This is an open-label study.

Patients receive oral sorafenib tosylate twice daily on days 1-28. Treatment repeats every 4 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients receive escalating doses of sorafenib tosylate (in the absence of grade 3 or 4 dose-limiting toxicity) until a pre-determined dose is reached.

Blood and urine samples are collected at baseline and periodically during study for VEGF level determination. Blood samples are analyzed for T4/T8, NK, CD25+, and Fox p3 by flow cytometry. Tumor tissue blocks or unstained slides are obtained for chemistry staining of VEGF.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

Inclusion Criteria:

* Histologically or cytologically confirmed renal cell carcinoma (RCC)

  * Must have a component of conventional clear cell RCC
  * Predominant clear cell component ≥ 75%
* Metastatic or unresectable disease (Measurable disease is defined as any lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as ≥ 20 mm by conventional techniques or ≥ 10 mm by spiral CT scan or MRI)
* Measurable or nonmeasurable disease, includes any of the following:

  * Small lesions, longest diameter < 20 mm by conventional techniques or < 10 mm by spiral CT scan
  * Bone lesions
  * Leptomeningeal disease
  * Ascites
  * Pleural/pericardial effusion
  * Lymphangitis cutis/pulmonitis
  * Abdominal masses that are not confirmed and followed by imaging techniques
  * Cystic lesions
  * Irradiated lesions, unless progression is documented after radiotherapy
* Paraffin RCC tissue blocks or unstained slides must be obtained for future chemistry staining of VEGF
* Karnofsky performance status 70-100%
* Fertile patients must use effective contraception (hormonal and/or barrier method) during and for 3 months after completion of study treatment
* Granulocyte count ≥ 1,500/µL
* Platelet count ≥ 100,000/µL
* AST/ALT ≤ 2.5 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 2.5 times ULN
* Serum bilirubin ≤ 1.5 times ULN
* Protein ≤ 1+ by urinalysis
* Creatinine ≤ 1.5 times ULN
* At least 4 weeks since prior major surgery and/or radiotherapy and recovered
* Prior palliative radiotherapy for metastatic lesion(s) allowed provided there is at least one measurable and/or evaluable lesion(s) that has not been irradiated
* More than 4 weeks since prior and no other concurrent anticancer therapy
* Concurrent continuation of bisphosphonates allowed for bone metastases prophylaxis

Exclusion Criteria:

* Patients with true papillary, sarcomatoid features without any clear cell component, chromophobe, oncocytoma, collecting duct tumors, or transitional cell carcinoma are not eligible
* No evidence of CNS metastases
* No imaging (MRI or CT scan of the brain) abnormality indicative of CNS metastases within past 42 days
* Not pregnant or nursing (negative pregnancy test)
* No ongoing hemoptysis
* No cerebrovascular accident within the past 12 months
* No peripheral vascular disease with claudication while walking less than 1 block
* No history of clinically significant bleeding
* No deep venous thrombosis or pulmonary embolus within the past year
* No significant cardiovascular disease, defined as NYHA class II-IV congestive heart failure, angina pectoris requiring nitrate therapy, or myocardial infarction within the past 6 months
* No uncontrolled hypertension, defined as systolic BP > 160 mm Hg and/or diastolic BP > 90 mm Hg while on medication
* No preexisting thyroid abnormality whose thyroid function cannot be maintained in the normal range by medication
* No uncontrolled psychiatric disorder
* No delayed healing of wounds, ulcers, and/or bone fractures
* No currently active second malignancy except nonmelanoma skin cancer (patients are not considered to have a 'currently active' malignancy if they have completed anticancer therapy and are considered by their physician to be at less than 30% risk of relapse)
* No more than one prior systemic therapy for RCC
* No prior vascular endothelial growth factor receptor agents
* No concurrent systemic corticosteroid therapy (except replacement therapy for adrenal insufficiency)

  o Topical and/or inhaled steroids allowed
* No concurrent full-dose oral or parenteral anticoagulation

  o Low-dose warfarin (1 mg) for maintenance of catheter patency or daily prophylactic aspirin allowed
* No concurrent Hypericum perforatum (St. John's wort)
* No concurrent ketoconazole, itraconazole, ritonavir, rifampin, or products containing grapefruit juice
* No concurrent hormonal therapy or chemotherapy o Concurrent hormones administered for non-disease related conditions (e.g., insulin for diabetes) allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2007-03-01 (Actual); Primary Completion 2009-10-31 (Actual); Study Completion 2014-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Hauke, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Sorafenib: The initial dose of Sorafenib will be administered orally with a dose of 400 mg twice a day, daily. Intrapatient dose escalation will occur as defined in the table below, providing no dose limiting toxicity (Grade 3 or 4) is observed. If grade 3 or 4 toxicity is observed, delay and dose modification will occur as defined in protocol. Once dose level 3 is reached, the patient will remain at that dose as defined in the protocol.
  Dose Level 1 Day 1-28 400 mg b.i.d. Dose Level 2 Day 29-56 600 mg b.i.d. Dose Level 3 Day 57- 800 mg b.i.d.
  A treatment cycle will be 4 weeks.
  Two 4-week cycles will be administered. At the completion of two cycles (week 8), restaging will occur. Patients will continue on therapy per study protocol.
Period: Overall Study
Arm/Group | Sorafenib
Started | 14
Completed | 11
Not Completed | 3

BASELINE CHARACTERISTICS:
Groups:
- Sorafenib: sorafenib tosylate: initial dose of Sorafenib will be administered orally with a dose of 400 mg twice a day, daily.Intrapatient dose escalation will occur providing no dose limiting toxicity (Grade 3 or 4) is observed. Dose level 2 600mg. Dose level 2 800mg
  flow cytometry: 15 ml of blood drawn for flow cytometry of T4/T8, NK, CD25+, and Fox p3 testing obtained at baseline and on days 28, 56, 84, and 112
  laboratory biomarker analysis: 15 ml of plasma and urine for storage and future determination of VEGF concentration will be obtained at baseline.10 ml of plasma and urine for storage and future determination of VEGF concentration will be obtained on days 28, 56, 84 and 112
Arm/Group | Sorafenib
Number analyzed (Participants) | 14
Age, Customized [Count of Participants; unit: Participants]
  Patients greater than or equal to 19 years of age | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Toxicity of Intrapatient Dose Escalation of Sorafenib Tosylate
Description: To evaluate the toxicity of dose escalating sorafenib, an estimation of the percentage of patients who are unable to tolerate those escalated doses will be made. Patients will be dose escalated every 4 weeks until a maximum dose of 800 mg BID is reached.
Time Frame: Study completion
Population: Evaluation of this data is not possible as the investigator performing the analysis has left the study center prior to completing the analysis and data was not provided.
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

2. Secondary Outcome: Response Rate
Description: The proportion of subjects with an objective response of complete or partial based on the RECIST Criteria
Time Frame: from the start of the treatment until disease progression/recurrence
Population: as for outcome 1
Arm/Group | Sorafenib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events and serious adverse events will be collected and reported on the forms beginning with the first dose of investigational product and continuing through the end of the study. (approximately 4 months)
Arm/Group | Sorafenib
All-Cause Mortality (participants affected / at risk) | 6/14
Serious Adverse Events (participants affected / at risk) | 2/14
Other Adverse Events (participants affected / at risk) | 11/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=14)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, weakness (General disorders) | 1 (1)
Other, shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, extremities tingling, numbness (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sorafenib (N=14)
Other- rash (Skin and subcutaneous tissue disorders) | 4 (7) — face
Other, pain (General disorders) | 5 (8)
Other, hand foot syndrome (Skin and subcutaneous tissue disorders) | 7 (7)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 6 (6)
Insomnia (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 8 (10)
Alopecia (Skin and subcutaneous tissue disorders) | 4 (4)
Other, upset stomach (Gastrointestinal disorders) | 1 (2)
Ejection fraction decreased (Investigations) | 1 (1)
Fatigue (General disorders) | 5 (9)
Retinal detachment (Eye disorders) | 1 (1)
Weight loss (Investigations) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 3 (3)
Gastroparesis (Gastrointestinal disorders) | 2 (2)
Other, mouth sensitivity (General disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 3 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 3 (3)
Other, elevated cardiac enzymes (Cardiac disorders) | 1 (1)
Other, stomach cramps (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Other, cramping (General disorders) | 2 (3)
Other, DVT (Vascular disorders) | 1 (1) — left leg
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, increased alkaline phosphatase (Investigations) | 1 (1)
Other, blood in stool (Gastrointestinal disorders) | 1 (1)
Other, weak urine stream (Investigations) | 1 (1)
Other, pale face (Investigations) | 1 (1)
Other, Bleeding gums (Infections and infestations) | 1 (1)
Other, hematemesis (Gastrointestinal disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Other, pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, soreness mouth and throat (Gastrointestinal disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Other, Blisters (Skin and subcutaneous tissue disorders) | 1 (2) — hands, foot
Other, pulmonary embolus (Vascular disorders) | 1 (1)
Other, renal insufficiency (Renal and urinary disorders) | 1 (1)
Other, tingling hands (Skin and subcutaneous tissue disorders) | 1 (1)
Other, lesions (Skin and subcutaneous tissue disorders) | 1 (1)
Other, swelling (Vascular disorders) | 2 (2) — hands and feet, left leg
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Other, Weakness (General disorders) | 1 (1)
Other, cracking, erythema fingertips (Skin and subcutaneous tissue disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Other, Hematochezia (Gastrointestinal disorders) | 1 (1)
Other, Soreness (Musculoskeletal and connective tissue disorders) | 1 (1) — extremities
Other, Tenderness/burning scalp (Skin and subcutaneous tissue disorders) | 1 (1)
Other, Neuropathy (Nervous system disorders) | 1 (1)
Other, Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Other, Stomatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Hematuria (trace) (Renal and urinary disorders) | 1 (1)
Other, decreased ionized calcium level (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Other, decreased magnesium level (Investigations) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Other, Leukoplakia (Infections and infestations) | 1 (1) — oral

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No